CLINICAL TRIAL: NCT06567197
Title: Multiple Sclerosis Treatment With Autologous Hematopoietic Stem Cell Transplantation (MS-ACT): A Long-term Prospective Observational Study in the Netherlands
Brief Title: Multiple Sclerosis Treatment With Autologous Hematopoietic Stem Cell Transplantation in the Netherlands
Acronym: MS-ACT
Status: Recruiting | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Joep Killestein, Clinical Professor, Amsterdam UMC, location VUmc
Other Study IDs: NL83783.018.23
Record Dates: First submitted 2024-06-25; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to study the long-term effects of autologous hematopoietic stem cell transplantation (aHSCT) in people with highly active relapsing-remitting multiple sclerosis. The study will evaluate the following items:

1. Disease activity
2. Safety and tolerability of aHSCT
3. Changes in the immune system

Participants will be subjected to frequent visits for five years after treatment with aHSCT. During these visits, clinical testing, evaluation by questionnaires, MRI scans and blood sampling will be performed.

ELIGIBILITY:
Inclusion Criteria:

* All patients approved for treatment with aHSCT in the Netherlands in accordance with the Dutch criteria for aHSCT treatment for RRMS

Exclusion Criteria:

* Contra-indications for treatment with aHSCT such as known hypersensitivity to the medication used for aHSCT
* Clinically relevant comorbidities preventing safe use of medication used for aHSCT
* Severe clinical depression
* Active addiction to drugs or alcohol
* Active infections such as but not limited to tuberculosis, cytomegalovirus, Epstein-Barr virus, herpes simplex, varicella zoster, viral hepatitis, toxoplasmosis, HIV or syphilis.
* Active malignancy or history of malignancy with the exception of local basal cell carcinoma or carcinoma in situ of the cervix

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with highly active relapsing-remitting multiple sclerosis are eligible for treatment with aHSCT in the Netherlands if they meet the criteria as defined by the Dutch National Health Care Institute.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Treatment efficacy | 2 years
  The proportion of patients with ne evidence of disease activity-3 (NEDA-3) as defined by: no clinical relapse, no disability progression, no radiological disease activity.

SECONDARY OUTCOMES:
Annual relapse rate | 2 years
Time to first relapse | 2 years
Confirmed disability progression (CDP) | 2 years
  Measured by the Expanded Disability Status Scale (EDSS) CDP-EDSS is defined as an increase of one point in the EDSS score from baseline to month 24.
Confirmed disability improvement (CDI) | 2 years
  Measured by the Expanded Disability Status Scale (EDSS) CDI-EDSS is defined as a decrease of one point in the EDSS score from baseline to month 24, with an absence of relapse at the point of assessment.
Progression independent of relapse activity (PIRA) | 2 years
  Defined as an episode of CDP without relapse during the 90 days before EDSS increase and during the 6-month period between the EDSS increase and the confirmation of disability progression.
Changes on the multiple sclerosis functional composite (MSFC) | 2 years
  MSFC consists of the timed 25-foot walk test, 9-hole peg test and standard digit modalities test (SDMT)
Brain/spinal cord MRI | 2 years
  Presence and number of contrast-enhancing lesions at baseline and the development of new or enlarging lesions between baseline and follow-up will be assessed.
Optical coherence tomography (OCT) | 2 years
  Developments of optic neuritis and longitudinal changes of the retinal nerve fiber layer will be assessed.
Side-effects and toxicity | 2 years
  Frequency and type of (serious) adverse events such as infections, secondary auto-immunity, fertility problems, clinical relevant changes on physical examination and use of concomitant medications will be assessed
Multiple Sclerosis Impact Scale-29 (MSIS-29) | 2 years
  Patient reported outcome measures about the impact of MS on daily life
EuroQoL 5D (EQ-5D-5L) | 2 years
  Patient reported outcome measures about quality of life
Modified Fatigue Impact Scale (MFIS-5) | 2 years
  Patient reported outcome measures about fatigue
Hospital Anxiety and Depression Scale (HADS) | 2 years
  Patient reported outcome measures about anxiety and depression
iMTA Medical Cost Questionnaire (iMCQ) | 2 years
  Patient reported outcome measures about medical consumption
iMTA Productivity Cost Questionnaire (iPCQ) | 2 years
  Patient reported outcome measures about productivity
Treatment Satisfaction Questionnaire for Medication (TSQM) | 2 years
  Patient reported outcome measures about medication
Biomarkers | 2 years
  Serum NfL and GFAP over time
Proteomics | 2 years
  Olink discover panel
Immune phenotyping | 2 years
  Characterization of innate and adaptive immune subsets with mass spectrometry imaging
Genetic analysis | 2 years
  Immune gene profiling for gene signatures predictive for response to aHSCT

CONTACTS AND LOCATIONS:
Overall Officials: J. Killestein, MSc, PhD, Principal Investigator — Amsterdam UMC
Locations (2):
- Netherlands (2):
  - Amsterdam UMC, Amsterdam
  - St. Antonius Hospital, Nieuwegein

IPD SHARING:
Plan to Share IPD: Undecided